CLINICAL TRIAL: NCT05755165
Title: Reducing Depression-related Stigma and Increasing Help-seeking Intentions: a Randomized Trial of Video Ads on Instagram
Brief Title: Adolescent Depression: Video Ads on Instagram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000028980_e; No NIH funding (Other: 12.06.23)
Record Dates: First submitted 2023-02-15; First posted 2023-03-06 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Depression; Stigmatization
MeSH Terms: conditions — Depression; Stereotyping

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Depression (Active Comparator): Adolescent depression
  Interventions: Behavioral: Depression
- Depression, adjusted (Active Comparator): Adolescent depression, impacted by racism
  Interventions: Behavioral: Depression, adjusted
- Control (Active Comparator): Control condition
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Depression — ~90-second selfie video of an adolescent discussing her history of depression, treatment, and recovery
  Arms: Depression
Behavioral: Depression, adjusted — ~90-second selfie video of an adolescent discussing her history of depression, treatment, and recovery - and including explicit reference to the role of anti-Black racism as a contributing factor
  Arms: Depression, adjusted
Behavioral: Control — ~90-second selfie video of an adolescent discussing everyday activities and interests, with no reference to depression or racism.
  Arms: Control

SUMMARY:
The purposes of this study are to test among adolescent viewers the utility of different types of selfie short video-based messaging to:

1. Reduce stigma and self-stigma related to depression, and
2. Increase treatment-seeking intentions.

DETAILED DESCRIPTION:
Intervention videos will each be self-recorded videos (of ~90-second duration) featuring the same underage professional (ages 16) acting as simulated participant. The investigators will post three brief videos ('video Ads') to achieve similar exposure among Instagram users, 14-18-year-old. The videos are: (a) depression video; (b) depression video adjusted to race experiences, and (c) control videos. All videos will feature by the same Black adolescent girl.

The investigators intend to assign ~10,000 individuals aged 14-18 in a randomized way, in equal proportions, and stratified by sex and race, to view one of the three videos.

Outcomes will include:

1. Primary outcome: engagement (a composite of likes, shares, comments, and views)
2. Secondary outcome: clicks on a designated link at the end of the video ad.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Living in the US
* Ages 14 - 18

Exclusion Criteria:

* None

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1235 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Engagement composite | Day 1: within 10 minutes of viewing the ad
  A sum of views, likes, shares, and comments on Instagram.
  The composite is an ordinal number ranging from 0 to n; higher values indicate greater engagement with the Instagram add.

SECONDARY OUTCOMES:
Clicks on designated link | Day 1: within 10 minutes of viewing the ad
  The number of clicks on a designated link at the end of the video ad.
  Clicks are an ordinal number ranging from 0 to n; higher values indicate greater engagement with the Instagram add.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Yale Child Center, New Haven, Connecticut
  - Yale Child Study Center, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin A, Calhoun A, Paez J, Amsalem D. Destigmatizing perceptions about Black adolescent depression: randomized controlled trial of brief social contact-based video interventions. J Child Psychol Psychiatry. 2022 Nov;63(11):1270-1278. doi: 10.1111/jcpp.13570. Epub 2022 Jan 23. PMID 35066880
- [Background] Amsalem D, Martin A. Reducing depression-related stigma and increasing treatment seeking among adolescents: randomized controlled trial of a brief video intervention. J Child Psychol Psychiatry. 2022 Feb;63(2):210-217. doi: 10.1111/jcpp.13427. Epub 2021 Apr 6. PMID 33821507
- [Background] Amsalem D, Halloran J, Penque B, Celentano J, Martin A. Effect of a Brief Social Contact Video on Transphobia and Depression-Related Stigma Among Adolescents: A Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e220376. doi: 10.1001/jamanetworkopen.2022.0376. PMID 35212749